CLINICAL TRIAL: NCT05149651
Title: Clinical and Radiographic Outcomes of Pulpotomy of Primary Molars Using Totalfill® Bioceramic Root Repair Material -Fast Set Putty, and ProRoot White MTA®. A Randomized Controlled Trial
Brief Title: Efficacy of Totalfill® and ProRoot MTA® as Pulpotomy Agent in Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC UZG 2016/0723 - 2016/0724
Record Dates: First submitted 2018-05-11; First posted 2021-12-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Extensively Decayed Primary Molars
Keywords: Totalfill; MTA; Bioactive; calcium silicate cement; Pulpotomy; Primary molars; Bioceramics
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Intervention Model Description: An experimental prospective double-blind, randomized clinical trial (RCT) with parallel design.
Who Masked: Participant, Outcomes Assessor
Masking Description: The included teeth were assigned randomly into two groups (Totalfill or MTA) using randomized sequences generated by the computer using Random Integer Generator (RANDOM.ORG, Randomness and Integrity Services Ltd.). The allocation ratio to the groups was set to be equal.
  To ensure double blinding at both patients and evaluators level during treatment, the type of material was concealed from the patient, and the patient had no information which material was used. In addition, the type of material was not mentioned in the patient file. Instead, it was replaced by a 4 digit code. The operators were also blinded for the type of material during the whole procedure starting from tooth preparation till the hemostasis was achieved and then were only informed at the time of material placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Totalfill (Experimental): Totalfill® Bioceramic Root Repair Material -Fast Set Putty used as pulpotomy agent to treat extensive decayed tooth indicated for pulpotomy
  Interventions: Drug: Totalfill
- MTA (Active Comparator): ProRoot White MTA® used as pulpotomy agent to treat extensive decayed tooth indicated for pulpotomy
  Interventions: Drug: MTA

INTERVENTIONS:
Drug: Totalfill — Totalfill® Bioceramic Root Repair Material -Fast Set Putty is a pre-mixed, bioactive calcium silicate cement which used as pulpotomy agent to treat extensive decayed tooth indicated for pulpotomy.
  Other Names: Totalfill® Bioceramic Root Repair Material -Fast Set Putty
  Arms: Totalfill
Drug: MTA — ProRoot White MTA® is a bioactive calcium silicate cement which used as pulpotomy agent to treat extensive decayed tooth indicated for pulpotomy.
  Other Names: ProRoot White MTA®
  Arms: MTA

SUMMARY:
An experimental prospective double-blind, randomized clinical trial (RCT) with parallel design. To evaluate the outcome of using 2 pulpotomy agents: Totalfill® as study group and mineral trioxide aggregate (MTA®) as a control.

DETAILED DESCRIPTION:
When a tooth decay is too deep and extended into the tooth pulp, then the tooth is not indicated to be treated with a filling. Therefore, removing the diseased pulp and then cover the rest with a suitable material is required. The Purpose of this study is to check the success of pulp treatment on deciduous molars with deep caries using 2 pulp treatment agents: (Totalfill® and MTA®). The use between the materials is randomly assigned. However, the use of the materials has no side effect or complications as it is a routine dental procedure.

The participants are healthy children aged between 3 and 9 years old, and the study is taking place in Ghent University Hospital, Ghent, Belgium, and it is planned to be conducted in duration of 4 years, which include 20 months for participants recruitment.

After placing the material, the tooth is restored with stainless steel crowns, and the participant was asked for follow up to check the tooth and to take dental x-ray every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient inclusion criteria

   * ASA 1 patient, Patient is a completely healthy & fit. No allergy or medical conditions.
   * Patient is indicated for treatment under General Anesthesia: young age, uncooperative and extensive treatment plan.
   * Parent agreed to participate in the study, and signed the written consent.
   * Patient attended the out-patients pediatric dental clinic in UZ Gent.
2. Tooth inclusion criteria 2.1. Clinical inclusion criteria:

   * Vital primary molars (first or second) with deep caries cavity with pulpal exposure.
   * Only mandibular primary molar were included
   * No spontaneous pain
   * No history of swelling
   * No sinus tract/ fistula
   * Absent of tenderness in percussion
   * No pathological mobility
   * Restorable tooth (stainless steel crown can be placed)
   * Hemostasis can be achieved with a dry cotton pellet after removal of Coronal pulp.

2.2. Radiographical inclusion criteria:

* At least 2/3rd of root is present
* Absence of internal or external root resorption
* Absence of pathologic root resorption
* Absence of periapical or furcation radiolucency

Exclusion Criteria:

If one or more of the criteria mentioned above is not fulfilled, the teeth were excluded from the study.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation | 6 months follow-up
  Success or failure of the pulpotomy treated teeth is scored based on the Clinical scoring criteria adapted from Zurn & Seale (2008). Score 1 and 2 was estimated as success, while 3 and 4 was estimated as failure.
Clinical evaluation | 12 months follow-up
  Success or failure of the pulpotomy treated teeth is scored based on the Clinical scoring criteria adapted from Zurn & Seale (2008). Score 1 and 2 was estimated as success, while 3 and 4 was estimated as failure.
Radiographic evaluation | 6 months follow-up
  Success or failure of the pulpotomy treated teeth is scored based on the Radiographic scoring criteria adapted from Zurn & Seale (2008). Score 1 and 2 was estimated as success, while 3 and 4 was estimated as failure.
Radiographic evaluation | 12 months follow-up
  Success or failure of the pulpotomy treated teeth is scored based on the Radiographic scoring criteria adapted from Zurn & Seale (2008). Score 1 and 2 was estimated as success, while 3 and 4 was estimated as failure.

SECONDARY OUTCOMES:
Time needed to place the material | Immediately after each intervention for a maximum of the intervention
  To measure the time consumed to place each material and then to compare them if there is a significant difference. After removing the coronal pulp and achieving the hemostasis . The operator start the timer when he places the material till restoring the tooth with GIC.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data will be available in the literature in the manuscript after publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication